CLINICAL TRIAL: NCT00017784
Title: Open-Label Safety Study of Valganciclovir in Patients With CMV Retinitis and AIDS Who Have Complications Due to IV Treatment
Brief Title: Valganciclovir in Patients With CMV Retinitis and AIDS Who Cannot Take Drugs by Injection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 268C; ML16356
Record Dates: First submitted 2001-06-11; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-06

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Infusions, Intravenous; Antiviral Agents; Cytomegalovirus Retinitis; valganciclovir
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; AIDS-Related Opportunistic Infections | interventions — Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir

SUMMARY:
The purpose of this study is to make valganciclovir available, before it is approved for marketing, to HIV-infected patients who have cytomegalovirus (CMV) retinitis (eye infection) and cannot take drugs by injection. This study also will look at the safety of using valganciclovir as starting and/or ongoing therapy.

CMV can cause serious AIDS-related infections in patients with HIV. Drugs that are effective against CMV eye infections can be given only by injection; this calls for a thin tube to be placed into a vein in the chest so that the patient is not put through getting too many needle sticks. An experimental drug, valganciclovir, is similar to 1 of these approved drugs, ganciclovir, but is more convenient and easier to use since it can be taken by mouth. Once in the body, valganciclovir changes to ganciclovir. Studies have shown that valganciclovir tablets can result in the same level of ganciclovir in the blood as ganciclovir injection.

DETAILED DESCRIPTION:
CMV causes sight- or life-threatening opportunistic infections in people with AIDS. Intravenous agents including ganciclovir, foscarnet, and cidofovir are presently approved as treatments for CMV retinitis within this population. Ganciclovir and foscarnet induction and maintenance therapy require daily infusions and usually require the use of long-term indwelling central venous catheters. Although the treatment interval of cidofovir is longer, administration necessitates the use of pre-hydration and probenecid in order to avoid a risk of renal toxicity. Oral ganciclovir is an alternative to the intravenous formulation for the maintenance treatment of CMV retinitis. However, because blood levels achieved after oral ganciclovir are low compared to intravenous, oral ganciclovir cannot be used for induction therapy. In an attempt to improve the bioavailability of ganciclovir, valganciclovir was developed. Valganciclovir is a ganciclovir prodrug which, when administered orally, is rapidly converted to the active compound ganciclovir during a first-pass process, with the majority of hydrolysis occurring pre-systemically. Studies have shown that valganciclovir tablets allow systemic exposure of ganciclovir comparable to that achieved with recommended doses of intravenous ganciclovir.

Patients undergo an ophthalmologic exam by an ophthalmologist and safety and other laboratory tests to establish eligibility. No specific visits are requested by the drug usage plan following enrollment; however, patients should be seen for safety and/or clinical assessments and medication dispensation at periodic visits, consistent with standard of care. An ophthalmologic exam should be performed again at Week 3 (no later than Week 4), at the end of the induction treatment phase consistent with standard of care in order to ensure adequate response to therapy. Valganciclovir is provided on a monthly basis and only as long as the patient is assessed and information provided in a timely manner. This supply will be terminated 1 month subsequent to when the drug is available by prescription, unless otherwise decided.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are 18 years of age or older.
* Are HIV-positive.
* Have active CMV retinitis, shown by an eye exam by an eye doctor, that needs treatment.
* Have had problems when drugs were given by injection, such as difficulty in finding a vein or problems (blood clots, vein inflammation, or infection) caused by injection devices.
* Agree to use effective methods of birth control (i.e., barrier methods) during the study and for 90 days after taking the study drug. Females who can have children must have a negative pregnancy test before entering the study.
* Stop breast-feeding before starting the study drug.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are pregnant or breast-feeding.
* Have developed CMV retinitis after a transplant.
* Have kidney disease and need hemodialysis.
* Are taking part in another drug study, unless approved by the study doctor.
* Take experimental drugs, or have taken them within 30 days before study entry, unless approved by the study doctor.
* Take drugs not allowed on the study, including foscarnet, cidofovir, and probenecid.
* Are not able to follow study procedures, including visits to the eye doctor and the study doctor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500

CONTACTS AND LOCATIONS:
Locations (9):
- United States (8):
  - Retina - Vitreous Associates Med Group, Beverly Hills, California
  - Wilbert Jordan, Paramount, California
  - Quest Clinical Research, San Francisco, California
  - Santa Clara Valley Med Ctr, San Jose, California
  - IDC Research Initiative, Altamonte Springs, Florida
  - Ingenix Kern McNeill Decatur, Atlanta, Georgia
  - Nashville Health Management Foundation / Vanderbilt Univ, Nashville, Tennessee
  - North Texas Infectious Disease Consultants, Dallas, Texas
- Fundacion Gastroenterologia de Diego, San Juan, Puerto Rico